CLINICAL TRIAL: NCT04409002
Title: A Phase II Study of Niraparib and Dostarlimab With Radiation in Patients With Metastatic Pancreatic Cancer
Brief Title: Niraparib + Dostarlimab + RT in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, Julie Koenig, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-538
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — niraparib; dostarlimab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib+Dostarlimab + Radiation (Experimental): Each study treatment cycle lasts 21 days
  * Niraparib oral, once a day, predetermined dose.Dosing will commence on cycle 1 day 1 and will continue until the participant is taken off treatment
  * Dostarlimab by intravenous infusion once every cycle for as long as they remain on the study
  * Radiation therapy on every other week day of cycle 2 only. Radiation will begin on Cycle 2 Day 1
  Interventions: Drug: Niraparib; Drug: Dostarlimab; Radiation: Radiation

INTERVENTIONS:
Drug: Niraparib — Niraparib oral, once a day, predetermined dose.Dosing will commence on cycle 1 day 1 and will continue until the participant is taken off treatment
  Other Names: Zejula
Drug: Dostarlimab — Dostarlimab by intravenous infusion once every cycle for as long as they remain on the study
Radiation: Radiation — Radiation therapy on every other week day of cycle 2 only. Radiation will begin on Cycle 2 Day 1

SUMMARY:
This research is being done to see how the combination of dostarlimab, niraparib, and radiation therapy works in controlling metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This two-stage single arm phase II trial will evaluate the efficacy of niraparib with dostarlimab and radiation therapy in patients with metastatic pancreatic cancer

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The names of the experimental interventions involved in this study are:

* Dostarlimab
* Niraparib
* Radiation Therapy

It is expected that about 25 people will take part in this research study. An initial 15 participants will be enrolled during the first stage and evaluated for treatment disease control, if none of the initial 15 participants achieve disease control the study will be terminated.

It is expected participants will be on the research study for as long as the experimental interventions are safe, and their metastatic pancreatic cancer does not progress with up to 5 years of follow up after participants stop taking the experimental interventions.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The U.S. Food and Drug Administration (FDA) has not approved dostarlimab as a treatment for any disease. Dostarlimab is a type of antibody (a protein that attaches to other cells to fight off infection) that is believed to work by attaching to a protein called PD-1 on Tcells.

This PD-1 protein controls parts of the immune system (the system in the body that fights off infections and diseases) by shutting down certain immune responses responsible for recognizing and destroying cancer cells. The investigators believe that dostarlimab will inhibit the PD-1 protein, thus allowing the immune cells to recognize and destroy cancer cells. The FDA has not approved niraparib for metastatic pancreatic cancer, but it has been approved for other uses. Niraparib is a type of drug called a "PARP inhibitor", which blocks DNA (the genetic material of cells) damage from being repaired or may prevent damage from occurring in the first place. In cancer treatment, inhibiting PARP may help kill cancer cells by not allowing the cancer cells to repair its DNA damage or prevent DNA damage from occurring. It is believed that the combination of dostarlimab, niraparib, and radiation therapy may have a greater effect on metastatic pancreatic cancer cells than when these interventions are used alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of pancreatic origin.
* Age > 18 years.
* ECOG performance status ≤ 1.
* Life expectancy of greater than 3 months.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥ 2,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * hemoglobin ≥ 9 g/dL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal(subjects with liver metastases can have an AST (SGOT) ≤ 5 x ULN
  * creatinine ≤ 1.5 x ULN OR
  * creatinine clearance* ≥ 60 mL/min (if using the Cockcroft-Gault formula)
  * total bilirubin ≤ 1.5 x ULN (subjects with Gilbert Syndrome can have a total bilirubin < 3 x ULN)
  * INR, PT, aPTT ≤ 1.5 x ULN (subjects receiving anticoagulant therapy must have PT or PTT within therapeutic range) *Creatinine clearance should be calculated per the following: CrCl (mL/min) = (140 - age [years]) x weight [kg] x 1.23 (x 0.85 if female)/ Serum creatinine (micromol/L)
* Women of childbearing potential (WoCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to initiating protocol therapy.

Non childbearing potential is defined as follows (by other than medical reasons):

* ≥45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 150 days after the last dose of study treatment. See Section 4.4 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.

  * Women of childbearing potential must agree to use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 6 months (30 days plus the time required for niraparib to undergo five half-lives/150 days) after the last dose of investigational drug.
  * Women must not be breastfeeding during the study or for 150 days after the last dose of investigational drug.
  * Men who are sexually active with WoCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving protocol therapy and who are sexually active with WoCBP will be instructed to adhere to contraception for a period of 6 months (150 days) after the last dose of investigational product. (Women who are not of childbearing potential, i.e. are postmenopausal as defined in the eligibility criteria or surgically sterile, as well as azoospermic men do not require contraception.) Ability to understand and the willingness to sign a written informed consent document
  * If applicable, stable dose of dexamethasone of 10mg or less for 4 weeks prior to initiation of investigational protocol therapy. Regimen must be completed >14 days prior to treatment start.
  * One previously unirradiated lesion amenable to radiotherapy at a dose of 8 Gy x 3 and can meet dose constraints, and another unirradiated measurable lesion > 1 cm in size outside the radiation field that can be used as measurable disease.
  * Patients must have had at least one line of prior treatment. Any prior line of treatment is permitted, including adjuvant.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded:

* Systemic anticancer or biological therapy including prior chemotherapy, immunotherapy, targeted small molecule therapy within 14 days prior to investigational agent, or those who have not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Participants with ≤ grade 2 neuropathy are an exception to these criteria and may qualify for the study. If the participant received major surgery, then they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Received investigational therapy ≥ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
* Major surgery ≤ 3 weeks prior to initiating protocol therapy and/or not recovered from any surgical effects.
* Received radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to day 1 of protocol therapy.
* Received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy
* Received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy. Known history of Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Active, known or suspected autoimmune disease that has required systemic treatment within the past 2 years other than vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants are permitted to use topical, ocular, intraarticular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Known history of active TB (Bacillus Tuberculosis). Testing is not required for eligibility purposes.
* Known hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. Testing is not required for eligibility purposes.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). These participants are at increased risk of lethal infections when treated with marrow suppressive therapy. Testing is not required for eligibility purposes.
* Known ≥ Grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent (within 90 days) myocardial infarction or psychiatric illness/social situations that would limit compliance with study requirements.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Known additional malignancy diagnosed, detected or treated ≤ 2 years prior to initiation of protocol therapy . Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known history of, or any evidence of active, non-infectious pneumonitis or interstitial lung disease.
* Active infection requiring systemic therapy
* Has received a live vaccine within 30 days of planned start of study therapy. Note:

Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Known hypersensitivity to niraparib and dostarlimab components or excipients.
* History of severe hypersensitivity reaction to any monoclonal antibody
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

Further imaging is not required for eligibility purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Koenig, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Niraparib+Dostarlimab + Radiation: Each study treatment cycle lasts 21 days
  * Niraparib oral, once a day, predetermined dose.Dosing will commence on cycle 1 day 1 and will continue until the participant is taken off treatment
  * Dostarlimab by intravenous infusion once every cycle for as long as they remain on the study
  * Radiation therapy on every other week day of cycle 2 only. Radiation will begin on Cycle 2 Day 1
  Niraparib: Niraparib oral, once a day, predetermined dose.Dosing will commence on cycle 1 day 1 and will continue until the participant is taken off treatment
  Dostarlimab: Dostarlimab by intravenous infusion once every cycle for as long as they remain on the study
  Radiation: Radiation therapy on every other week day of cycle 2 only. Radiation will begin on Cycle 2 Day 1
Period: Overall Study
Arm/Group | Niraparib+Dostarlimab + Radiation
Started | 18
Completed | 15
Not Completed | 3
Not completed — Disease progression prior to starting study treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  Age 30-39 years | 2
  Age 40-49 years | 1
  Age 50-59 years | 5
  Age 60-69 years | 7
  Age 70-79 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate With RECIST 1.1 Criteria
Description: Disease control rate (DCR) is the percentage of participants who experienced a complete response (CR), partial response (PR), or stable disease (SD) assessed by the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria below.
  * CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * PR = At least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum diameters.
  * SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the baseline sum diameters while on study.
  * Progressive Disease (PD) = At least 20% increase in the sum of longest diameters of target lesions, taking as reference the baseline sum diameters while on study. Appearance of one or more new lesions is also considered progression.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 15
Participants | 0

2. Secondary Outcome: Disease Control Rate With irRECIST Criteria
Description: Disease control rate (DCR) is the percentage of participants who experienced a immune-related complete response (irCR), partial response (irPR), or stable disease (irSD) assessed by the Immune-Related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria below.
  * irCR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * irPR = At least 30% decrease in the sum of longest diameters of target lesions, compared to baseline.
  * irSD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, compared to baseline.
  * Immune-related Progressive Disease (irPD) = At least 20% increase in the sum of longest diameters of target lesions AND at least 5mm absolute increase, compared to baseline. Appearance of one or more new lesions is also considered progression. Confirmation scan required at least 4 weeks later.
Time Frame: up to 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time duration from the first day of protocol treatment to the earlier date of disease progression or death due to any cause. PFS time will be censored at the date of last follow-up for surviving patients with disease control.
Time Frame: up to 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 15
months | 1.6 [1.1 to 2.7]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time duration from the first day of protocol treatment to the date of death due to any cause, and will be censored at the date of last follow-up for patients still alive.
Time Frame: up to 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 15
months | 3.1 [1.5 to 7.7]

5. Secondary Outcome: Number of Treatment-Related Adverse Events Per CTCAE v5.0
Description: Treatment-related adverse events (TRAEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, as grades 3-5 and at least possibly attributed to study treatment. TRAEs are evaluated from the start of study treatment through 30-days after the last treatment dose.
Time Frame: up to 19 weeks
Measure: Number; unit: treatment-related adverse events
Arm/Group | Niraparib+Dostarlimab + Radiation
Number analyzed (Participants) | 15
treatment-related adverse events
  Grade 3 TRAEs | 17
  Grade 4 TRAEs | 3
  Grade 5 TRAEs | 0

ADVERSE EVENTS:
Time Frame: up to 17 months
Description: Adverse event evaluations per CTCAE v5.0
Arm/Group | Niraparib+Dostarlimab + Radiation
All-Cause Mortality (participants affected / at risk) | 14/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib+Dostarlimab + Radiation (N=15)
Fever (General disorders) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib+Dostarlimab + Radiation (N=15)
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 11
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 7
Aortic valve disease (Cardiac disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 4
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bacteremia (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 2
Blood bilirubin increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac troponin T increased (Investigations) | 2
CD4 lymphocytes decreased (Investigations) | 10
Chills (General disorders) | 4
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Dysuria (Renal and urinary disorders) | 2
Edema limbs (General disorders) | 5
Encephalopathy (Nervous system disorders) | 1
Endocarditis infective (Infections and infestations) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — blood in the corner of right eye. no pain. no change in vision
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 12
Fever (General disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — radiation induced proctitis
Gastrointestinal pain (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Glucosuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Insomnia (Psychiatric disorders) | 2
Lethargy (Nervous system disorders) | 1
Localized edema (General disorders) | 2
Lymphocyte count decreased (Investigations) | 3
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myocarditis (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Primary malignant neoplasm of endometrium
Neutrophil count decreased (Investigations) | 2
Obesity (Metabolism and nutrition disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Palpitations (Cardiac disorders) | 2
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 6
Platelet count decreased (Investigations) | 8
Portal vein thrombosis (Hepatobiliary disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 — Breast Cancer
Restlessness (Psychiatric disorders) | 1
Scleral disorder (Eye disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 5
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Stroke (Nervous system disorders) | 1
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 7
Thrush (Infections and infestations) | 2
Thyroid stimulating hormone increased (Investigations) | 1
Tremor (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 3
Vaginal dryness (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 4

LIMITATIONS AND CAVEATS:
A two-stage design was used, requiring disease control in at least one of the first 15 patients before proceeding to the full accrual of 25 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04409002/Prot_SAP_000.pdf